CLINICAL TRIAL: NCT00009906
Title: Phase III Randomized, Intergroup Trial Assessing the Clinical Activity Of STI-571 at Two Dose Levels in Patients With Unresectable or Metastatic Gastrointestinal Stromal Tumors (GIST) Expressing the Kit Receptor Tyrosine Kinase (CD117)
Brief Title: Comparison of Two Different Doses of STI571 in Treating Patients With Metastatic or Unresectable Gastrointestinal Stromal Tumor
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Eastern Cooperative Oncology Group (Network); SWOG Cancer Research Network (Network); NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-02372; NCI-2012-02372 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S0033; INT-S0033; CDR0000068422; CAN-NCIC-S0033; CLB-80004; SWOG-S0033; E-S0033; S0033 (Other: SWOG); S0033 (Other: CTEP); U10CA180888 (NIH); U10CA032102 (NIH); N01CM17003 (NIH)
Record Dates: First submitted 2001-02-02; First posted 2004-02-03 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-06

CONDITIONS: Gastrointestinal Stromal Tumor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (imatinib mesylate) (Experimental): Patients receive oral imatinib mesylate once daily.
  Interventions: Drug: Imatinib Mesylate
- Arm II (imatinib mesylate) (Experimental): Patients receive oral imatinib mesylate twice daily.
  Interventions: Drug: Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib Mesylate — Given orally

SUMMARY:
Randomized phase III trial to compare the effectiveness of two different doses of STI571 in treating patients who have metastatic or unresectable gastrointestinal stromal tumor. STI571 may interfere with the growth of tumor cells and may be an effective treatment for cancer. It is not yet known which dose of STI571 is more effective in treating gastrointestinal stromal tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the overall and progression-free survival of patients with CD117-expressing metastatic or unresectable gastrointestinal stromal tumor treated with two different doses of imatinib mesylate.

II. Compare the confirmed, unconfirmed, complete, and partial response rates in patients treated with these regimens.

III. Compare the toxic effects of these regimens in these patients.

OUTLINE: This is a randomized study. Patients are randomized to one of two treatment arms.

Arm I: Patients receive oral imatinib mesylate once daily.

Arm II: Patients receive oral imatinib mesylate twice daily.

Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients in arm I with progressive disease may cross over to arm II and receive treatment in the absence of further disease progression.

Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 600 patients will be accrued for this study within 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a biopsy proven diagnosis of gastrointestinal stromal tumor (GIST) which is distantly metastatic or unresectable; tumors must meet BOTH of the following criteria:

  * The primary must be of visceral or intra-abdominal origin
  * All patients must have immunohistochemical documentation of KIT (CD117) expression by tumor documented by DAKO antibody staining for suggested methodology) Material must be submitted to the CALGB Pathology Coordinating Center for pathology review; it is strongly recommended that snap-frozen tissue biopsy and sera be stored for future submission whenever possible
* Patient must have measurable or non-measurable disease by conventional scan imaging (CT or MRI) or physical examination; tests used to assess disease must have been performed within 28 days prior to registration; if a target lesion has been previously embolized or irradiated, there must be objective evidence of progression to be considered for response assessment
* Patient must have an identified team (including a medical oncologist and a surgeon) to provide care
* Patient must not have known brain metastasis
* Patient must have a Zubrod performance status of 0 - 3
* Patient must have resolution of transient toxicities from any prior therapy to =< grade 1 (NCI-CTC version 2.0)
* The patient must not have received chemotherapy, biologic therapy or any other investigational drug for any reason within 28 days prior to registration; patients must not have had a major surgery within 14 days prior to registration
* If day 14 or 28 falls on a weekend or holiday, the limit may be extended to the next working day

  * In calculating days of tests and measurements, the day a test or measurement is done is considered day 0; therefore, if a test is done on a Monday, the Monday two weeks later would be considered day 14; this allows for efficient patient scheduling without exceeding the guidelines
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* At the time of patient registration, the treating institution's name and ID number must be provided to the Data Operations Center in Seattle in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered into the data base
* Patients on lower dose arm (Arm 1) will be allowed to increase the daily dose of STI-571 in the case of disease progression; if there is questionable disease progression, the treating investigator should contact the primary Study Coordinator, Dr. George Demetri at 617/632-3985 to review progression information and discuss treatment options

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 748 (Actual)
Dates: Start 2000-12; Primary Completion 2007-05 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to 3 years
Progression-free survival | From date of registration to date of first observation of progressive disease or death due to any cause, assessed up to 3 years
Toxicity defined as any grade 3 or greater organ toxicity, or any grade 4 or greater hematological toxicity as assessed by CTCAE version 2.0 | Up to 3 year after completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: George Demetri, Principal Investigator — SWOG Cancer Research Network
Locations (144):
- United States (132):
  - Western Regional CCOP, Phoenix, Arizona
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Highlands Oncology Group-Rogers, Rogers, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Long Beach Community Hospital, Long Beach, California
  - University of Southern California/Norris Cancer Center, Los Angeles, California
  - University of California at Los Angeles Health System, Los Angeles, California
  - Sutter Cancer Research Consortium, Novato, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - University of California San Diego, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Santa Rosa Memorial Hospital, Sana Rosa, California
  - Stanford University Hospitals and Clinics, Stanford, California
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Middlesex Hospital, Middletown, Connecticut
  - MedStar Oncology Network, Washington D.C., District of Columbia
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Hematology Oncology Associates, Lake Worth, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Jesse Brown Veterans Affairs Medical Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Central Illinois CCOP, Decatur, Illinois
  - Alexian Brothers Medical and Cancer Center, Elk Grove Village, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Mid-Illinois Hematology Oncology Associates, Normal, Illinois
  - Advocate Lutheran General Hospital., Park Ridge, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kansas City CCOP, Prairie Village, Kansas
  - Stormont-Vail Regional Health Center, Topeka, Kansas
  - Our Lady Bellefonte Hospital, Ashland, Kentucky
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Michigan Cancer Research Consortium Community Clinical Oncology Program, Ann Arbor, Michigan
  - University of Michigan University Hospital, Ann Arbor, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - Unity Hospital, Fridley, Minnesota
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Joseph's Health Center, Saint Charles, Missouri
  - Ozark Health Ventures LLC-Cancer Research for The Ozarks Springfield, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical CCOP, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Winthrop University Hospital, Mineola, New York
  - Beth Israel Medical Center, New York, New York
  - New York University Langone Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeast Cancer Control Consortium CCOP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus CCOP, Columbus, Ohio
  - Dayton CCOP, Dayton, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Sky Lakes Medical Center - Cancer Treatment Center, Klamath Falls, Oregon
  - Western Oncology Research Consortium, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Salem Hospital, Salem, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Aria Health-Torresdale Campus, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Upstate Carolina CCOP, Spartanburg, South Carolina
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Central Vermont Medical Center, Barre, Vermont
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - Rutland Regional Medical Center, Rutland, Vermont
  - Virginia Oncology Associates-Hampton, Hampton, Virginia
  - Virginia Mason CCOP, Seattle, Washington
  - Group Health, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Northwest CCOP, Tacoma, Washington
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
- Canada (10):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Hamilton and District Urology Association McMaster Institute, Hamilton, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Health Research Institute-General Division, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University Department of Oncology, Montreal, Quebec
- Puerto Rico (2):
  - San Juan Veterans Affairs Medical Center, San Juan
  - San Juan City Hospital, San Juan

REFERENCES:
- [Derived] Heinrich MC, Rankin C, Blanke CD, Demetri GD, Borden EC, Ryan CW, von Mehren M, Blackstein ME, Priebat DA, Tap WD, Maki RG, Corless CL, Fletcher JA, Owzar K, Crowley JJ, Benjamin RS, Baker LH. Correlation of Long-term Results of Imatinib in Advanced Gastrointestinal Stromal Tumors With Next-Generation Sequencing Results: Analysis of Phase 3 SWOG Intergroup Trial S0033. JAMA Oncol. 2017 Jul 1;3(7):944-952. doi: 10.1001/jamaoncol.2016.6728. PMID 28196207